CLINICAL TRIAL: NCT02160223
Title: Sugammadex Compared With Neostigmin/Atropin for Neuromuscular Block Reversal in Patients With Obstructive Sleep Apnea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, DILEK YAZICIOGLU, Dr, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Sugammadex-OSA
Record Dates: First submitted 2014-06-08; First posted 2014-06-10 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2012-01

CONDITIONS: Obstructive Sleep Apnea
Keywords: sugammadex; neostigmine; obstructive sleep apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugammadex (Experimental): Group S patients will receive 2 mg kg -1 sugammadex at the end of surgery
  Interventions: Drug: Sugammadex
- Neostigmine (Active Comparator): Group N patients will receive 50 µg kg-1 neostigmine and 05 mg atropin at the end of surgery
  Interventions: Drug: Neostigmine

INTERVENTIONS:
Drug: Sugammadex — Group S patients will receive 2 mg kg -1 sugammadex at he end of surgery
  Arms: Sugammadex
Drug: Neostigmine — Patient in Gropu N will receive 50 µg kg-1 neostigmin and 05 mg atropin at the end of surgery
  Arms: Neostigmine

SUMMARY:
Incomplete recovery of neuromuscular function after surgery can lead to respiratory complications. Patients with obstructive sleep apnea (OSA) are prone to respiratory complications after surgery. Neostigmin and sugammadex are used for neuromuscular reversal.

The aim of this study was to compare sugammadex and neostigmin regarding efficacy, incidence of respiratory complications and cost in patients undergoing surgery for OSA

DETAILED DESCRIPTION:
This prospective double blind controlled study will be conducted after obtaining informed written patient consent.

Simple randomization will be accomplished with a computer-generated sequence of numbers and sealed envelopes will be used to allocate patients into 2 groups.

Group N will receive 50 µg kg-1 neostigmin,+05 mg atropin Group S will receive sugammadex 2mg kg-1 sugammadex at the and of surgery. Patients will enter the operation room without receiving premedication Heart rate, noninvasive blood pressures, body temperature, BIS, end-tidal respiratory gases and neuromuscular function (acceleromyography) will be monitored Propofol will be used for anesthesia induction Rocuronium 0.6 mg kg-1 will be used to facilitate intubation Anesthesia will be maintained with sevoflurane in oxygen and nitrous oxide, BIS will be maintainen between 40-60 Additional rocuronium doses will be administered when the TOF T2 is observed At the end of surgery, volatile anesthesia will be discontinued, the study drug will be administered according to group allocation and the TOF response at this time will be recorded Time to obtain TOF0.9 will be recorded Time to extubation, time to recovery, time spent in the operation room will be recorded Respiratory and cardiovascular complications (bradycardia, tachycardia, hypertention, ritmia, bronchospasm, laringospasm, breath holding, cough, desaturation, hypoxia, NIMV, reintubation) and treatments during anesthesia emergence will be recorded Patients will be transfered to the PACU, time spent in PACU and respiratory and cardiovascular complications (bradycardia, tachycardia, hypertention, ritmia, bronchospasm, laringospasm, breath holding, cough, desaturation, hypoxia, NIMV, reintubation) and treatments during PACU stay will be recorded After achieving an Aldrete score >9 patients will be transfered to the ward. Patients who can not achieve Aldrete score >9 after 1 hour will be transfered to the ICU.

Respiratory and cardiovascular complications and treatments in the ICU will be recored

ELIGIBILITY:
Inclusion Criteria:

ASA I-III Schedulled for surgery for obstructive sleep apnea -

Exclusion Criteria:

Neurouscular disorders hepatic or renal dysfunction allergy to study drugs using medication that could interfere with NMBAs pregnancy breasth feeding

-

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
TOF0.9 time | postoperative 5 minutes
  TOF 0.9 time will be recorded form the TOF watch after the study drug administration

SECONDARY OUTCOMES:
desaturation | postoperative 5 minutes
  patients will be monitored for desaturation after extubation
bradycardia | postoperative 5 minutes
  heart rate will bw monitored after extubation
tachycardia | postoperative 5 minutes
  heart rate will be monitored after extubation

OTHER OUTCOMES:
operation room time | postoperative 30 minutes
  the time elapsed from the study drug administration to the the time the patient was transfered to the PACU
PACU time | poastoperative 1 hour
  time elapsed from the the patient entering the PACU to the time the patient left the PACU

CONTACTS AND LOCATIONS:
Overall Officials: Dilek yazicioglu, Dr, Principal Investigator — Dişkapı yildirim beyazit Teaching and Research Hospital
Locations (1):
- Diskapi Yildirim Beyazit Teaching and Research Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Jones RK, Caldwell JE, Brull SJ, Soto RG. Reversal of profound rocuronium-induced blockade with sugammadex: a randomized comparison with neostigmine. Anesthesiology. 2008 Nov;109(5):816-24. doi: 10.1097/ALN.0b013e31818a3fee. PMID 18946293
- [Background] Khuenl-Brady KS, Wattwil M, Vanacker BF, Lora-Tamayo JI, Rietbergen H, Alvarez-Gomez JA. Sugammadex provides faster reversal of vecuronium-induced neuromuscular blockade compared with neostigmine: a multicenter, randomized, controlled trial. Anesth Analg. 2010 Jan 1;110(1):64-73. doi: 10.1213/ane.0b013e3181ac53c3. Epub 2009 Aug 27. PMID 19713265
- [Background] Kaw R, Pasupuleti V, Walker E, Ramaswamy A, Foldvary-Schafer N. Postoperative complications in patients with obstructive sleep apnea. Chest. 2012 Feb;141(2):436-441. doi: 10.1378/chest.11-0283. Epub 2011 Aug 25. PMID 21868464